CLINICAL TRIAL: NCT04369339
Title: Immediate Colposcopy Findings Among Women With High Risk HPV Other Than HPV 16/18 and Normal Cytology
Brief Title: Colposcopy Findings Among Women With High Risk HPV Other Than HPV 16/18 and Normal Cytology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Serdar Aydın, Assoc. Prof., Bezmialem Vakif University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OHRHPVCOLP
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Human Papillomavirus Infection
Keywords: Human Papilloma Virus; negative for intraepithelial lesions or malignancy; HPV16; HPV18
MeSH Terms: conditions — Papillomavirus Infections; Neoplasms | interventions — Colposcopy

STUDY DESIGN:
Intervention Model Description: prospective cohort study comparing the immediate colposcopy findings among women with HrHPV other than HVPV16/18 and negative cytology
Who Masked: Outcomes Assessor
Masking Description: outcomes assessor blind to clinical data and cytology results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Other High Risk HPV Positivity (Experimental): Colposcopy performed to women with High risk HPV positive ,negative for intraepithelial lesions or malignancy cytology
  Interventions: Other: Colposcopy
- HPV16/18 (Active Comparator): Colposcopy performed to women with HPV 16/18 positive ,negative for intraepithelial lesions or malignancy cytology
  Interventions: Other: Colposcopy

INTERVENTIONS:
Other: Colposcopy

SUMMARY:
Abnormal cervical cytology was the most common reason for women being referred to the colposcopy unit. We prospectively included the women with negative cytology (negative for intraepithelial lesions or malignancy (NILM)) and positive High RiskHPV test other than HPV 16 or HPV 18. Comparing the immediate colposcopy findings among women with High Risk HPV other than HVPV16/18 and negative cytology and determine positive predictive values for CIN2+ of other high risk HPV genotypes

ELIGIBILITY:
Inclusion Criteria:

* negative cytology (negative for intraepithelial lesions or malignancy (NILM)) and positive HrHPV test other than HPV 16 or HPV 18

Exclusion Criteria:

* Previous diagnosis for cervical cancer Previous diagnosis for vaginal cancer Previous diagnosis for cervical dysplasia Previous diagnosis for ASCUS previous history of cervical conisation or hysterectomy previous history ofhysterectomy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Dysplasia | 1 month
  Pathologic diagnosis of cervical dysplasia

IPD SHARING:
Plan to Share IPD: No